CLINICAL TRIAL: NCT07285109
Title: The Impact of Qualia Vitamin C+ on Blood Vitamin C Levels
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qualia Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: QLS-020
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Vitamin C Deficiency
MeSH Terms: conditions — Ascorbic Acid Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qualia Vitamin c+ (Active Comparator): Qualia Vitamin C+ manufactured by Qualia Life Sciences
  Interventions: Dietary Supplement: Qualia Vitamin C+
- Placebo (Placebo Comparator): Rice flour placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Qualia Vitamin C+ — Qualia Vitamin C+ manufactured by Qualia Life Sciences
  Arms: Qualia Vitamin c+
Dietary Supplement: Placebo — Rice flour
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group, study evaluating the effect of a Qualia Vitamin C+ formulation on Whole Blood Vitamin C levels in the blood of healthy adults aged 25 years or older. Approximately 36 participants will be randomized to one of two study arms: Qualia Vitamin C+ or placebo. Each participant will take two capsules of their assigned product once daily in the morning, with or without food, over a 28-day period. The primary outcome is the change in blood vitamin C levels, assessed via in lab blood collection at baseline and study completion. Secondary endpoints include questionnaires measuring health-related cognitive functioning and stress (PROMIS Cognitive Function - Short Form 8a and the Perceived Stress Scale-10), the Single-item Assessment of Immune Fitness, evaluation of safety and tolerability, and an Overall Experience Questionnaire (Appendices 1, 4-7). All assessments, including electronic questionnaires, are completed remotely without in-person visits.

ELIGIBILITY:
Inclusion criteria:

Provide voluntary, written, informed consent to participate in the study. Agree to provide a valid cell phone number and are willing to receive communications through text.

Can read and write English. Willing to complete questionnaires, records, and diaries associated with the study.

Healthy male and female participants aged 25 years or older. Willing to go to an Ulta Labs Patient Service Center location for a Blood Vitamin C Test (baseline and Day 29) and located within a convenient distance of participating locations. [Note: The services offered by Ulta Lab Tests are available only in the United States and not to residents of the states of New Jersey, New York, and Rhode Island.] Willing to avoid starting new or stopping any existing dietary supplements throughout the study.

Exclusion criteria:

Women who are pregnant, breastfeeding, or planning to become pregnant or start breastfeeding during the trial.

Known food intolerances/allergy to any ingredients in the product. Having any of the following conditions: Psychiatric conditions, neurologic disorders, endocrine disorders, cancer.

Having had a significant cardiovascular event in the past 6 months. Taking MAO inhibitors, SSRIs, or any other psychiatric or neurological medicines On immunosuppressive therapy. Adults lacking capacity to consent.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2026-02-11 (Estimated); Study Completion 2026-02-11 (Estimated)

PRIMARY OUTCOMES:
To assess between-group differences in the change in blood Vitamin C levels from baseline to Day 28 | 0-28 days
  To assess between-group differences in the change in blood Vitamin C levels from baseline to Day 28 following supplementation with Qualia Vitamin C+ versus placebo.

SECONDARY OUTCOMES:
To assess within-group and between-group differences in PROMIS Cognitive Function - Short Form 8a | baseline to day 14 and 28
To assess within-group and between-group differences in Perceived Stress Scale-10 domain scores | baseline to day 14 and 28
To assess within-group and between-group differences in Single-item Assessment of Immune Fitness | baseline to day 14 and 28
To assess within-group differences in the change in blood Vitamin C levels | baseline to day 28
To evaluate side effect profiles using a custom Safety and Tolerability survey | baseline to day 14 and 28

CONTACTS AND LOCATIONS:
Locations (1):
- Qualia Life Sciences, Carlsbad, California, United States

IPD SHARING:
Plan to Share IPD: No